CLINICAL TRIAL: NCT06715891
Title: A Multicenter, Double-blind, Placebo-controlled, Randomized, Parallel-group Clinical Trial of the Efficacy and Safety of Raphamin in the Treatment of Acute Respiratory Viral Infection in Children Aged 3-12 Years
Brief Title: Clinical Trial of the Efficacy and Safety of Raphamin in the Treatment of ARVI in Children Aged 3-12 Years
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMH-407-010
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Acute Respiratory Viral Infection
Keywords: respiratory viral infection; children; aged 3-12 years

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, randomized, parallel-group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Raphamin (Experimental): Per os without food. The tablet should be kept in mouth until completely dissolved.
  On day 1 of treatment, 8 tablets should be taken using the following regimen: 1 tablet every 30 minutes for the first 2 hours (5 tablets in total for 2 hours), then 1 more tablet 3 times at equal intervals during the same day. On day 2 and onwards, 1 tablet should be taken 3 times a day. The duration of treatment is 5 days.
  Interventions: Drug: Raphamin
- Placebo (Placebo Comparator): Placebo using the Raphamin dosage regimen.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Raphamin — Tablet for oral use.
  Other Names: MMH-407
  Arms: Raphamin
Drug: Placebo — Tablet for oral use.
  Arms: Placebo

SUMMARY:
Multicenter double-blind placebo-controlled randomized in parallel groups clinical trial.

DETAILED DESCRIPTION:
Design: a multicenter, double-blind, placebo-controlled, randomized, parallel-group clinical trial.

The trial will enroll outpatients of either gender aged 3 to 12 years with clinical manifestations of acute respiratory viral infection (ARVI) within the first 24 hours after the disease onset. Patient enrollment will be conducted in 2 stages during the seasonal incidence of ARVI. First, children aged 6-12 years will be enrolled in the trial. Once the required number of patients is reached, an "unblinded" interim analysis with the primary efficacy endpoint assessment and safety analysis will be performed. Based on the data from the unblinded interim analysis, a decision will be made whether the age range of enrollment can be expanded from 3 to 12 years. Patient enrollment will not be stopped until the results of the "unblinded" interim analysis are available.

After the parent/adopter signs the information sheet and informed consent form for the patient's parents/adopters to participate in the clinical trial, the medical history will be collected, thermometry, objective examination, laboratory tests will be performed, and concomitant therapy will be recorded. The severity of ARVI symptoms will be assessed using a 4-point scale.

The nasopharyngeal swabs for PCR diagnosis and verification of respiratory viruses will be performed prior to therapy to confirm the viral etiology of ARVI.

If a patient meets all inclusion criteria and does not have any exclusion criteria, at Visit 1 (Day 1), they will be randomized into one of two groups: Group 1 patients will receive Raphamin according to the dosage regimen for 5 days; Group 2 patients will receive Placebo using the Raphamin dosage regimen for 5 days.

The trial will utilize an electronic patient diary (EPD) where the patient will make daily records of morning and evening axillary body temperature (measured with a classic mercury-free thermometer) and symptoms of the disease (ARVI Symptom Severity Score). In addition, antipyretic dosing (if applicable) as well as any possible worsening of the patient's condition (if applicable, to assess safety / to record adverse events) will also be recorded in the patient diary. The investigator will instruct the parent/adopter on how to complete the diary. At Visit 1, the parent/adopter together with the physician will record the severity of ARVI symptoms and body temperature in the diary.

The patient will be observed for 14 days (screening, randomization - up to 1 day, treatment - 5 days, follow-up - up to 2 days; deferred "phone visit" - day 14).

During the treatment and follow-up period, patients/physicians will pay 3 visits, and the fourth "phone visit" will be scheduled additionally: 1) physician/patient visits - on days 1, 5 and 7 (Visits 1, 2 and 3) - at the health center or at home; 2) a phone "visit" by the physician (Visit 4) - on day 14.

During Visits 2 and 3, the physician will perform objective examination, record changes in the disease symptoms, concomitant therapy, and monitor the completion of the diary. During Visit 3, compliance will be assessed and laboratory tests will be performed.

A phone "visit" will be performed to interview the parent/adopter about the patient's condition, presence/absence of secondary bacterial/viral complications, and use of antibiotics.

Symptomatic therapy and therapy for concomitant diseases will be permitted during the trial except for the drugs listed under "Prohibited Concomitant Treatment".

ELIGIBILITY:
Inclusion Criteria:

1. Children of either gender aged 3 to12 years .
2. Diagnosis of ARVI based on the medical examination: axillary temperature ≥37.8°C at the time of examination + total severity of general symptom score ≥4 points, nasal/throat/chest symptoms ≥2 points (ARVI Symptom Severity Score).
3. 24 hours from the ARVI onset .
4. Availability of a patient information sheet and an informed consent form for the patient's parents/adopters for patient participation in the clinical trial signed by one parent/adopter of the patient.

Exclusion Criteria:

1. Clinical symptoms of severe influenza/ARVI requiring hospitalization.
2. Suspected pneumonia, bacterial infection (including otitis media, sinusitis, urinary tract infection, meningitis, sepsis, etc.) requiring the administration of antibiotics from the first day of disease.
3. Suspected early manifestations of diseases that have onset symptoms similar to those of ARVI (other infectious diseases, influenza-like syndrome at the onset of systemic connective tissue diseases and other pathologies).
4. Patients who require administration of antiviral medications that are prohibited for use in this trial.
5. History or prior diagnosis of primary and secondary immunodeficiency.
6. History/suspicion of oncology of any localization (except for benign neoplasms).
7. Exacerbation or decompensation of chronic diseases (diabetes mellitus, cerebral palsy, cystic fibrosis, primary ciliary dyskinesia, bronchopulmonary dysplasia, malformations of the respiratory and ENT organs, etc.) affecting the patient's ability to participate in the clinical trial.
8. Malabsorption syndrome, including congenital or acquired lactase or other disaccharidase deficiency, galactosemia.
9. Allergy/hypersensitivity to any component of the medicines used in the treatment.
10. Use of medications listed under "Prohibited Concomitant Treatment" within 2 weeks prior to inclusion in the trial.
11. Patients whose parents/adopters, from the investigator's point of view, will not comply with the observation requirements during the trial or follow the procedure for taking the test drugs.
12. History of mental illness of the patient (except for attention deficit hyperactivity disorder), parents/adopters of the patient.
13. Participation in other clinical trials within 3 months prior to inclusion in this trial.
14. A patient's parent/adopter is related to any of the on-site research personnel directly involved in the trial, or is the immediate family member of the investigator. 'Immediate family members' mean spouses, parents, children, or siblings, whether related or adopted.
15. The patient's parent/adopter is employed by OOO "NPF "MATERIA MEDICA HOLDING", i.e., is an employee of the company, a temporary contract employee, or a designated official responsible for conducting the trial or their immediate family member.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 374 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to resolution of ARVI symptoms (PCR-confirmed) | 14 days
  Time from recording the disease symptoms at Visit 1 until resolution of the disease symptoms.
  Resolution of ARVI symptoms will be defined if axillary temperature is ≤37.3°C for 24 hours (without further increase during observation period) + lack/presence of ARVI general symptoms ≤2 points. Based on the patient's diary.

SECONDARY OUTCOMES:
ARVI severity (clinically diagnosed, including PCR-confirmed) | From day 1 to day 6
  Вased on the area under curve (AUC) results for the total severity score. The total disease severity score will be calculated based on the severity of each of the ARVI symptoms (body temperature, general symptoms, and nasal/throat and chest symptoms in points). To calculate the total score, absolute values of body temperature measured in degrees Celsius will be converted into relative units (or points) based on the following classification: ≤37.3°C=0 points; 37.4-38.0°C=1 point; 38.1-39.0°C=2 points; ≥39.1°C =3 points.
Percentage of patients with resolution of ARVI symptoms | 14 days
  Clinically diagnosed, including PCR-confirmed. Based on medical records.
Time to resolution of ARVI symptoms | 14 days
  Clinically diagnosed, including PCR-confirmed. Based on medical records.
Percentage of patients with resolution of ARVI symptoms (PCR-confirmed) | 14 days
  Based on medical records.
Dosing frequency of antipyretics | From day 1 to day 3
  Based on the patient's diary.
Percentage of patients with worsening of the disease | From day 4 to day 14
  Development of complications requiring antibiotics or hospitalization.
Number of Participants With Adverse Events (AEs) | From day 1 to day 6
  Presence and nature of adverse events during therapy. Based on medical records.
Severity of AEs | From day 1 to day 6
  The intensity (severity) of adverse events. Based on medical records.
Causal Relationship of AEs to the Sudy Drug | From day 1 to day 6
  The causal relationship to the study drug of adverse events. Based on medical records.
Outcome of AEs | From day 1 to day 6
  The outcome of adverse events. Based on medical records.
Changes in Vital Signs (Blood Pressure) measured in mm Hg | On Visit 1 (day 1), Visit 2 (day 5) and Visit 3 (day 7)
  Blood Pressure measured in mm Hg. Based on medical records.
Changes in Vital Signs (Heart Rate) | On Visit 1 (day 1), Visit 2 (day 5) and Visit 3 (day 7)
  Pulse Rate measured in beats per minute. Based on medical records.
Changes in Vital Signs (Breathing Rate) | On Visit 1 (day 1), Visit 2 (day 5) and Visit 3 (day 7)
  Respiratory Rate measured in breaths per minute. Based on medical records.
Changes in Vital Signs (Axillary temperature) | On Visit 1 (day 1), Visit 2 (day 5) and Visit 3 (day 7)
  Temperature is measured in the armpit using a classic mercury-free thermometer. Based on medical records.
Percentage of Patients With Clinically Significant Abnormal Laboratory Tests | On Visit 1 (day 1) and Visit 2 (day 5)
  Measure is based on the Hematology, blood chemistry, and urinalysis parameters, which are beyond the reference values.

CONTACTS AND LOCATIONS:
Locations (29):
- Russia (29):
  - Gatchina Clinical Interdistrict Hospital, Gatchina
  - Kazan State Medical University/Department of Hospital Pediatrics, Kazan'
  - LLC "MedLight", Kazan'
  - Regional Clinical Hospital # 2, Krasnodar
  - Specialized Clinical Infectious Diseases Hospital, Krasnodar
  - Central Research Institute of Epidemiology/Clinical Department of Infectious Pathology, Moscow
  - Morozovskaya Children's City Clinical Hospital of the Moscow City Health Department, Moscow
  - First Moscow State Medical University named after I.M. Sechenov/Department of Childhood Diseases, Moscow
  - Llc "Diagnostics and Vaccines", Moscow
  - Novosibirsk State Medical University/Clinic "Medical Advisory Center", Novosibirsk
  - Omsk State Medical University/Department of Hospital Pediatrics with a Course of Continuing Professional Education, Omsk
  - City Children's Clinical Polyclinic # 5, Perm
  - LLC "Professor's Clinic", Perm
  - LLC "4D Ultrasound Clinic", Pyatigorsk
  - Clinical and diagnostic center "Health", Rostov-on-Don
  - Ryazan State Medical University named after Academician I.P. Pavlov/Department of Children's Diseases with a course in hospital pediatrics, Ryazan
  - Children's City Polyclinic # 44, Saint Petersburg
  - Saint Petersburg State Pediatric Medical University/Department of Infectious Diseases of Adults and Epidemiology, Saint Petersburg
  - Children's City Polyclinic # 35, Saint Petersburg
  - Samara Regional Children's Clinical Hospital named after N.N. Ivanovoy/Department of Medical Rehabilitation, Samara
  - Samara State Medical University/Department of Hospital Pediatrics, Samara
  - National Research Mordovian State University named after N.P. Ogarev/Department of Pediatrics/, Saransk
  - Saratov City Children's Clinical Hospital, Saratov
  - Smolensk State Medical University/Department of Children's Diseases of the Medical and Dental Faculties, Smolensk
  - Bashkir State Medical University/Department of Outpatient and Emergency Pediatrics, Ufa
  - Yaroslavl State Medical University/Department of Pediatrics, Institute of Continuous Professional Education, Yaroslavl
  - Clinical Hospital # 2, Yaroslavl
  - Children's City Clinical Hospital # 11 Ekaterinburg, Yekaterinburg
  - Ural State Medical University/Department of Infectious Diseases, Phthisiology and Pulmonology, Yekaterinburg

IPD SHARING:
Plan to Share IPD: No